CLINICAL TRIAL: NCT06608719
Title: Retrospective Study on the Safety and Therapeutic/Improvement Effects of Intravenous Administration of SHED-CM for ALS
Brief Title: Retrospective Study on the Safety and Therapeutic/Improvement Effects of Intravenous Administration of SHED-CM for ALS (SHED-CAH2023)
Status: Completed | Type: Observational
Sponsor: Hitonowa Medical (Other)
Responsible Party: Sponsor
Other Study IDs: SHED-CM-ALS-H-2023
Record Dates: First submitted 2024-07-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS - Amyotrophic Lateral Sclerosis; Stem Cells; Conditioned Medium; Therapy; Safety; Regenerative Medicine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Receiving the study drug: Patients diagnosed with ALS who visited our hospital and were administered SHED-CM between January 1, 2022, and November 30, 2023.
  Interventions: Biological: The study drug is SHED-CM manufactured by U-Factor

INTERVENTIONS:
Biological: The study drug is SHED-CM manufactured by U-Factor — Patients diagnosed with ALS were administered SHED-CM

SUMMARY:
In this study, we will retrospectively evaluate the safety and efficacy of administering SHED-CM for the treatment of ALS.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a progressive and irreversible neurodegenerative disease with limited treatment options. Advances in regenerative medicine have opened new avenues for therapeutic interventions. This retrospective cohort study evaluated the safety and efficacy of stem cells from human exfoliated deciduous teeth-conditioned media (SHED-CM) in 24 patients with ALS treated at a single facility between January 1, 2022, and November 30, 2023. Safety assessments included adverse events, vital signs, and laboratory test changes before and after administration, whereas efficacy was measured using the ALS Functional Rating Scale-Revised (ALSFRS-R), grip strength, and forced vital capacity. while ALSFRS-R scores typically decline over time, the progression rate in this cohort was slower, suggesting a potential delay in disease progression. Alternatively, improvements in muscle strength and mobility were observed in some patients. Although adverse events were reported in only 3% of cases (no serious allergic reactions), the treatment-induced changes in vital signs and laboratory results were not clinically significant. The SHED-CM treatment appears to be a safe and potentially effective therapeutic option for patients with ALS. Further research is needed to optimize the SHED-CM treatment; however, this study lays the groundwork for future exploration of regenerative therapies for ALS.

ELIGIBILITY:
Inclusion Criteria:

* patients who visited our clinic between January 1, 2022 and November 30, 2023 and have been diagnosed with ALS
* male and female patients aged between 16 and 90 years old
* ALSFRS-R score of 12 or more at the time of initial visit

Exclusion Criteria:

* Patients who have a tracheostomy at the time of visit.
* Patients who have expressed their refusal to participate in this study.

Ages: 38 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Amyotrophic Lateral Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
All Adverse Events | after the treatment
  This measure will check the total number of adverse events (AEs) reported during the study, categorized by CTCAE Ver 5.0 .
Number of Clinically Significant Changes in Laboratory Test Results | Baseline (pre-treatment) and after 4th treatment
  This measure will track the number of events where clinically significant abnormalities are detected in laboratory test parameters, including blood count, biochemistry, and coagulation function tests. Changes from baseline to after the 4th treatment session will be evaluated based on predefined clinical thresholds.
Number of Clinically Significant Changes in Vital Signs | Baseline (pre-treatment), post-treatment, and after 4th treatment
  This measure will evaluate the number of events where clinically significant changes in vital signs occur. Parameters include systolic blood pressure, diastolic blood pressure, pulse rate, body temperature, and SpO2. Each event will be assessed at two time points: immediately after treatment and after the 4th treatment session, comparing values to baseline.
Safety assessment during the study period: Adverse events - Self- and other findings | after the treatment
  Medical examination, subjective findings, Other findings

SECONDARY OUTCOMES:
Efficacy assessment: Changes in Amyotrophic Lateral Sclerosis Functional Rating Scale Revised version | Change from baseline at 16 weeks
  The revised ALS Functional Rating Scale in ALS Patients. This scale is scored from 0 to 48, the higher the score the better.
Efficacy assessment: Changes in %FVC | Change from baseline at 16 weeks
  % forced vital capacity in percent
Efficacy assessment: Changes in grip strength | Change from baseline at 16 weeks
  grip strength in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Hitonowa Medical, Chiyoda City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
This was a retrospective cohort study including patients diagnosed with ALS who visited our hospital between January 1, 2022, and November 30, 2023. We enrolled pa-tients with ALS who received SHED-CM within this period, had a score of 12 or higher on the ALS Functional Rating Scale-Revised (ALSFRS-R), and did not undergo trache-ostomy. All administered data were evaluated for safety. Several patients experienced difficulties presenting to the hospital due to the progression of their ALS; therefore, we evaluated the efficacy of the drug from the first to the 12th dose, which were adminis-tered consecutively, and for which all patients presented to the hospital.
Supporting Information: Study Protocol, CSR
Time Frame: The original data presented in the study are openly available without restrictions.
Access Criteria: The original data presented in the study are openly available in FigShare at 10.6084/m9.figshare.26201615.
URL: https://doi.org/10.6084/m9.figshare.26201615.v1

REFERENCES:
- [Background] Oki R, Izumi Y, Fujita K, Miyamoto R, Nodera H, Sato Y, Sakaguchi S, Nokihara H, Kanai K, Tsunemi T, Hattori N, Hatanaka Y, Sonoo M, Atsuta N, Sobue G, Shimizu T, Shibuya K, Ikeda K, Kano O, Nishinaka K, Kojima Y, Oda M, Komai K, Kikuchi H, Kohara N, Urushitani M, Nakayama Y, Ito H, Nagai M, Nishiyama K, Kuzume D, Shimohama S, Shimohata T, Abe K, Ishihara T, Onodera O, Isose S, Araki N, Morita M, Noda K, Toda T, Maruyama H, Furuya H, Teramukai S, Kagimura T, Noma K, Yanagawa H, Kuwabara S, Kaji R; Japan Early-Stage Trial of Ultrahigh-Dose Methylcobalamin for ALS (JETALS) Collaborators. Efficacy and Safety of Ultrahigh-Dose Methylcobalamin in Early-Stage Amyotrophic Lateral Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2022 Jun 1;79(6):575-583. doi: 10.1001/jamaneurol.2022.0901. PMID 35532908
- See also: We referenced this paper because of the Phase III trial in ALS. — http://pubmed.ncbi.nlm.nih.gov/35532908/